CLINICAL TRIAL: NCT02979353
Title: A Randomized Controlled Trial to Deprescribe for Older Patients With Polypharmacy Transferred From the Hospital to Skilled Nursing Facilities
Brief Title: A Randomized Controlled Trial to Deprescribe for Older Patients With Polypharmacy
Acronym: Shed-Meds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sandra Simmons, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01AG053264-01 (NIH); R01AG053264 (NIH)
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Polypharmacy; Care Transitions; Geriatric Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shed-Meds: A Patient-Centered Deprescribing Intervention (Experimental): Participants assigned to the intervention group will receive a clinical review of their prescribed medications by a research clinician (Pharmacist, Physician, and/or Nurse Practitioner) followed by a patient interview to assess their willingness to discontinue or reduce some of their medicines based on the clinical recommendations of the team. Hospital and out-patient providers also will be part of the deprescribing decision process. Deprescribing actions will be initiated in the hospital prior to discharge and continue through the skilled nursing facility stay.
  Interventions: Behavioral: Shed-Meds: A Patient-Centered Deprescribing Intervention
- Control Group (No Intervention): Participants assigned to the control group will receive usual care as it is normally provided by the hospital and skilled nursing facility treatment teams. Research staff will monitor their prescribed medications in both care settings but not make any recommendations or changes, unless a safety issue is identified.

INTERVENTIONS:
Behavioral: Shed-Meds: A Patient-Centered Deprescribing Intervention — The goal of the intervention is to safely deprescribe medications, as defined by dose reductions and stopped medications, based on a combination of clinical criteria and patient preferences.
  Arms: Shed-Meds: A Patient-Centered Deprescribing Intervention

SUMMARY:
This randomized, controlled trial will evaluate the effects of an intervention to reduce exposure to medications among hospitalized older adults discharged to skilled nursing facilities (SNFs). The goal of the intervention is to safely deprescribe medications, as defined by dose reductions and stopped medications, based on a combination of clinical criteria and patient preferences. The investigators will evaluate the effects of the intervention on the total number of medications prescribed to patients at hospital and SNF discharge and at home 90-days after SNF discharge along with the prevalence of eight geriatric syndromes, medication adherence, and health status.

DETAILED DESCRIPTION:
This randomized, controlled trial will evaluate the effects of an intervention to reduce exposure to medications among hospitalized older adults discharged to skilled nursing facilities (SNFs). This study will be conducted in one university-affiliated hospital and 14 area SNFs to enroll approximately 1,300 total participants across five project years. Patients discharged to SNF represent the largest segment of Medicare beneficiaries discharged to post-acute care services and are a particularly high risk group for loss of independence and other poor clinical outcomes. This investigative team recently completed a Centers for Medicare and Medicaid Services (CMS) Innovation Award, which provides strong preliminary data related to the prevalence of polypharmacy and the relationship between polypharmacy and geriatric syndromes (e.g., medications associated with falls) in this patient population. Based on these data, the investigators developed a structured deprescribing intervention protocol ("Shed-Meds") coupled with standardized screening assessments for eight geriatric syndromes to be implemented in the hospital and continued during the SNF stay. The goal of the intervention is to safely deprescribe medications, as defined by dose reductions and stopped medications, based on a combination of clinical criteria and patient preferences. This trial will evaluate the effects of this intervention on medication exposure, medication adherence, geriatric syndromes, and health status across the care transitions from hospital to SNF to home to include a 90-day follow-up period after SNF discharge. The overarching hypothesis is that reducing medications for older patients across the continuum of care will favorably impact geriatric syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at Vanderbilt University Medical Center
* Medicare-eligible
* Discharged from VUMC to a post acute care facility
* Has polypharmacy as defined by > 5 medications
* Able to self-consent or has a proxy (surrogate)
* Speaks English (due to interview-based assessments)
* Primary home residence within one of 9 surrounding counties (due to home visit during follow-up phase)

Exclusion Criteria:

* Resides in long-term care
* Is currently on hospice or otherwise has a limited life expectancy (< 6 months).
* Enrolled in a clinical drug trial
* Has Stage IV Cancer Diagnosis
* Incarcerated or homeless
* Unable to self-consent and does not have a surrogate

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra F Simmons, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be shared, per written request and completion of formal data sharing agreement approved by the institution

REFERENCES:
- [Background] Vasilevskis EE, Shah AS, Hollingsworth EK, Shotwell MS, Kripalani S, Mixon AS, Simmons SF. Deprescribing Medications Among Older Adults From End of Hospitalization Through Postacute Care: A Shed-MEDS Randomized Clinical Trial. JAMA Intern Med. 2023 Mar 1;183(3):223-231. doi: 10.1001/jamainternmed.2022.6545. PMID 36745422
- [Background] Kim JL, Lewallen KM, Hollingsworth EK, Shah AS, Simmons SF, Vasilevskis EE. Patient-Reported Barriers and Enablers to Deprescribing Recommendations During a Clinical Trial (Shed-MEDS). Gerontologist. 2023 Mar 21;63(3):523-533. doi: 10.1093/geront/gnac100. PMID 35881109
- [Background] Hollingsworth EK, Shah AS, Shotwell MS, Simmons SF, Vasilevskis EE. Older Patient and Surrogate Attitudes Toward Deprescribing During the Transition From Acute to Post-Acute Care. J Appl Gerontol. 2022 Mar;41(3):788-797. doi: 10.1177/07334648211015756. PMID 35164584
- [Background] Shah AS, Hollingsworth EK, Shotwell MS, Mixon AS, Simmons SF, Vasilevskis EE. Sources of medication omissions among hospitalized older adults with polypharmacy. J Am Geriatr Soc. 2022 Apr;70(4):1180-1189. doi: 10.1111/jgs.17629. Epub 2021 Dec 30. PMID 34967444
- [Result] Vasilevskis EE, Shah AS, Hollingsworth EK, Shotwell MS, Mixon AS, Bell SP, Kripalani S, Schnelle JF, Simmons SF; Shed-MEDS Team. A patient-centered deprescribing intervention for hospitalized older patients with polypharmacy: rationale and design of the Shed-MEDS randomized controlled trial. BMC Health Serv Res. 2019 Mar 14;19(1):165. doi: 10.1186/s12913-019-3995-3. PMID 30871561

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shed-Meds: A Patient-Centered Deprescribing Intervention | Control Group
Started | 186 | 186
Hospital Phase | 174 | 181
Post-Acute Care Phase | 142 | 142
7-Day Follow-Up | 137 | 133
60-Day Follow-Up | 128 | 125
Completed | 116 | 115
Not Completed | 70 | 71
Not completed — Hospital Discharge to Non-Partner PAC or Non- PAC Location | 24 | 29
Not completed — Withdrawal by Subject | 16 | 12
Not completed — Death | 10 | 11
Not completed — Transfer to Hospice Care | 19 | 14
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shed-Meds: A Patient-Centered Deprescribing Intervention | Control Group | Total
Number analyzed (Participants) | 186 | 186 | 372
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 76.4 [69.5 to 85.3] | 76.9 [66.9 to 84.6] | 76.8 [69.1 to 84.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 112 | 229
  Male | 69 | 74 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 186 | 182 | 368
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 30 | 57
  White | 158 | 155 | 313
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 186 | 186 | 372
Total Number of Medications at Enrollment [Median (Inter-Quartile Range); unit: Medications] | 24.0 [19.2 to 29.0] | 23.0 [19.0 to 29.0] | 23.0 [19.0 to 29.0]
Anticholinergic and Sedative Drug Burden Index [Median (Inter-Quartile Range); unit: score on a scale] — A Drug Burden Index (DBI) score is calculated for each anticholinergic and sedative medication by dividing the individual medication's prescribed daily dose by the sum of the minimum effective dose (per FDA minimum recommended dose) and the patient's daily dose. The score range for each individual medication is 0 to 1, and the Anticholinergic & Sedative DBI reported is the sum of the individual medication scores. The Anticholinergic & Sedative DBI has a minimum score of 0 and no maximum. Higher scores indicate a higher drug burden (i.e., lower score is a better outcome).
  score on a scale | 4.1 [2.9 to 5.4] | 4.5 [3.1 to 6.3] | 4.2 [2.9 to 5.8]
Vulnerable Elders Survey 13 (VES-13) [Median (Inter-Quartile Range); unit: score on a scale] — The Vulnerable Elders Survey 13 (VES-13) is a self-rating of functional health status, and it consists of 4 groups of questions: age, self-perceived health, difficulties to perform 6 specific activities, and difficulties to perform daily living tasks due to health concerns. The total score ranges from 0 to 10. A score >=3 was considered to show impairment (i.e., worse outcome). Population: The number analyzed differs from the overall group N due to missing or incomplete participant assessment data for this measure.
  score on a scale
    number analyzed (Participants) | 157 | 153 | 310
    (all) | 7 [3 to 8] | 7 [3 to 8] | 7 [3 to 8]
Adherence to Refills and Medications Scale (ARMS) [Median (Inter-Quartile Range); unit: score on a scale] — Trained research staff administered the Adherence to Refills and Medication Scale (ARMS). Participants indicate the extent of their adherence on a 4-point Likert-like scale. Responses range from 1="none of the time" to 4="all of the time," and are summed to produce an overall adherence score ranging from 12-48, with lower values indicating better adherence (better outcome). Population: The number analyzed differs from the overall group N due to missing or incomplete participant assessment data for this measure.
  score on a scale
    number analyzed (Participants) | 141 | 136 | 277
    (all) | 14 [13 to 16] | 15 [13 to 18] | 15 [13 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Medications
Description: The number of medications a participant is taking. This includes all prescribed and over-the-counter medications and both scheduled and as-needed (PRN) medications.
Time Frame: Hospital Discharge, Post-Acute Care Discharge, and 90 days after discharge from the PAC
Population: Outcomes are reported for three different study time points (Hospital Discharge, Post-Acute Care Discharge, and 90-Day Follow Up After PAC Discharge). Both the Intervention and Control groups experienced attrition at each time point. The "number analyzed" below for each time point reflects the number of participants who completed that particular study time point.
Measure: Median (Inter-Quartile Range); unit: Medications
Arm/Group | Shed-Meds: A Patient-Centered Deprescribing Intervention | Control Group
Number analyzed (Participants) | 174 | 181
Medications
  Hospital Discharge (approximately 3 days after study enrollment) | 15 [12 to 18] | 16 [12 to 19]
  Post-Acute Care Discharge (approximately 31 days after study enrollment): number analyzed (Participants) | 142 | 142
  Post-Acute Care Discharge (approximately 31 days after study enrollment) | 13 [10 to 16] | 15 [12 to 19]
  90 Day Follow-Up After PAC Discharge (approximately 122 days after study enrollment): number analyzed (Participants) | 116 | 115
  90 Day Follow-Up After PAC Discharge (approximately 122 days after study enrollment) | 12 [9 to 16] | 14 [11 to 18]
Statistical Analysis 1: Comparison: Shed-Meds: A Patient-Centered Deprescribing Intervention vs Control Group; Statistical Analysis 1 applies to the Hospital Discharge timepoint (average 3 days after study enrollment); Test type: Superiority; p = 0.017, Mixed Models Analysis; Risk Ratio (RR) = 0.96
Statistical Analysis 2: Comparison: Shed-Meds: A Patient-Centered Deprescribing Intervention vs Control Group; Statistical Analysis 2 applies to the Post-Acute Care Discharge time point (occurred on average 31 days after study enrollment); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Risk Ratio (RR) = 0.86
Statistical Analysis 3: Comparison: Shed-Meds: A Patient-Centered Deprescribing Intervention vs Control Group; Statistical Analysis 3 applies to the 90 Day Follow-Up After PAC Discharge (occurred, on average, 122 days after study enrollment); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Risk Ratio (RR) = 0.85

2. Secondary Outcome: Total Drug Burden Index (DBI): Anticholinergic and Sedative Drug
Description: A Drug Burden Index (DBI) score is calculated for each anticholinergic and sedative medication by dividing the individual medication's prescribed daily dose by the sum of the minimum effective dose (per FDA minimum recommended dose) and the patient's daily dose. The score range for each individual medication is 0 to 1, and the Anticholinergic & Sedative DBI reported is the sum of the individual medication scores. The Anticholinergic & Sedative DBI has a minimum score of 0 and no maximum. Higher scores indicate a higher drug burden (i.e., lower score is a better outcome).
Time Frame: Hospital Discharge, Post-Acute Care Discharge, and 90 days after discharge from PAC
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Shed-Meds: A Patient-Centered Deprescribing Intervention | Control Group
Number analyzed (Participants) | 174 | 181
score on a scale
  Hospital Discharge (approximately 3 days after study enrollment) | 2.4 [1.5 to 3.4] | 2.9 [1.9 to 4.1]
  Post-Acute Care Discharge (approximately 31 days after study enrollment): number analyzed (Participants) | 142 | 142
  Post-Acute Care Discharge (approximately 31 days after study enrollment) | 2.2 [1.3 to 3.1] | 2.7 [1.5 to 4.3]
  90-Day Follow-Up After PAC Discharge (approximately 122 days after study enrollment): number analyzed (Participants) | 116 | 115
  90-Day Follow-Up After PAC Discharge (approximately 122 days after study enrollment) | 2.0 [1.0 to 2.8] | 2.3 [1.3 to 3.7]
Statistical Analysis 1: Comparison: Shed-Meds: A Patient-Centered Deprescribing Intervention vs Control Group; Statistical Analysis 1 applies to the Hospital Discharge time point (occurred, on average, 3 days after study enrollment); Test type: Superiority; p = 0.02, Regression, Linear; Mean Difference (Net) = -0.28
Statistical Analysis 2: Comparison: Shed-Meds: A Patient-Centered Deprescribing Intervention vs Control Group; Statistical Analysis 2 applies to Post-Acute Care Discharge time point (occurred, on average, 31 days after study enrollment); Test type: Superiority; p < 0.00001, Regression, Linear; Mean Difference (Net) = -0.59
Statistical Analysis 3: Comparison: Shed-Meds: A Patient-Centered Deprescribing Intervention vs Control Group; Statistical Analysis 3 applies to 90-Day Follow Up After PAC Discharge time point (occurred, on average, 122 after study enrollment); Test type: Superiority; p = 0.01, Regression, Linear; Mean Difference (Net) = -0.35

ADVERSE EVENTS:
Time Frame: All adverse events including all-cause mortality and serious adverse events were continuously monitored from participant enrollment through final follow-up timepoint at 90-days following post-acute care discharge, up to 295 days.
Description: The study used NIH/NIA definitions for adverse and serious adverse events. Serious adverse events included escalation of care to the intensive care unit (during baseline hospitalization), rehospitalization (after baseline), and death. Data for all unplanned healthcare utilizations and death are reported here regardless of cause or study-relatedness.
Arm/Group | Shed-Meds: A Patient-Centered Deprescribing Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 10/186 | 11/186
Serious Adverse Events (participants affected / at risk) | 59/186 | 76/186
Other Adverse Events (participants affected / at risk) | 12/186 | 7/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shed-Meds: A Patient-Centered Deprescribing Intervention (N=186) | Control Group (N=186)
Heart Failure (Cardiac disorders) | 6 (9) | 11 (11)
Pneumonia (Infections and infestations) | 8 (8) | 6 (7)
Cardiac Arrhythmias (Cardiac disorders) | 8 (8) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (9)
Urinary Tract Infections (Infections and infestations) | 5 (7) | 6 (11)
Infections - Pathogen Unspecified (Infections and infestations) | 4 (4) | 6 (6)
Bacterial Infections Disorders (Infections and infestations) | 3 (5) | 6 (8)
Renal Disorders (Renal and urinary disorders) | 3 (3) | 4 (4)
Vascular Hypotensive Disorders (Vascular disorders) | 2 (2) | 5 (5)
Encephalopathy (Nervous system disorders) | 1 (1) | 5 (5)
Sepsis - Pathogen unspecified (Infections and infestations) | 3 (4) | 3 (3)
Bone & Joint Fractures (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Central Nervous System Vascular Disorders (Nervous system disorders) | 4 (7) | 1 (2)
General System Disorders (NEC) (General disorders) | 1 (1) | 4 (4)
Coronary Artery Disorder (Cardiac disorders) | 1 (1) | 3 (3)
Gastrointestinal Motility and Defecation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Seizures (Nervous system disorders) | 1 (1) | 3 (3)
Bronchial Disorders (excludes neoplasms) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Electrolyte and Fluid Balance Conditions (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mental Disorders (Psychiatric disorders) | 1 (1) | 2 (2)
Cerebral Injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Depressive Disorders (Psychiatric disorders) | 0 (0) | 2 (2)
Exocrine Pancreas Conditions (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Signs & Symptoms (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal Stenosis & Obstructions (Gastrointestinal disorders) | 2 (2) | 0 (0)
Glucose Metabolism Disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vascular Hypertensive Disorders (Vascular disorders) | 0 (0) | 2 (3)
Anaemias (NEC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anxiety Disorders & Symptoms (Psychiatric disorders) | 0 (0) | 1 (1)
Calcium Metabolic Disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Delusion Symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
Device Issues (General disorders) | 1 (1) | 0 (0)
Embolism & Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Fungal Infection Disorders (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder Disorders (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haematology Investigations (Investigations) | 0 (0) | 1 (1)
Joint Disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Male Reproductive Tract Infections & Inflammations (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Peripheral Neuropathies (Nervous system disorders) | 0 (0) | 1 (1)
Phosphorous Metabolism Disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Plasma Cell Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Poisoning & Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Related Injuries & Complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary Hypertensions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Spleen Disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary Tract Signs & Symptoms (Renal and urinary disorders) | 0 (0) | 1 (1)
Vascular Haemorrhagic Disorders (Vascular disorders) | 0 (0) | 1 (1)
Viral Infectious Disorders (Infections and infestations) | 0 (0) | 1 (1) — COVID-19
White Blood Cell Disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shed-Meds: A Patient-Centered Deprescribing Intervention (N=186) | Control Group (N=186)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Mental Status Changes (Psychiatric disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT02979353/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT02979353/ICF_000.pdf